CLINICAL TRIAL: NCT03130361
Title: Evaluation of the Impact of a Wearable Noninvasive Positive Pressure Ventilation Device on Physical Activity and Quality of Life in Patients With COPD
Brief Title: Wearable Noninvasive Positive Pressure Ventilation Device in COPD
Acronym: VITABREATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icadom (Industry)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-A01297-44
Record Dates: First submitted 2016-08-16; First posted 2017-04-26 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Non-Invasive Ventilation
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Noninvasive ventilation (Experimental): Participants will use the device at home by intermittence during or after physical activities for reducing dyspnea or for shortening dyspnea-recovery time over a 4-week period.
  Interventions: Device: Non-Invasive Ventilation

INTERVENTIONS:
Device: Non-Invasive Ventilation

SUMMARY:
The objective is to assess the impact of a wearable Noninvasive Positive Pressure Ventilation, on physical activity and quality of life in patients with severe COPD, complaining of dyspnea.

DETAILED DESCRIPTION:
In order to avoid the occurrence of uncomfortable dyspnea, patients with Chronic Obstructive Pulmonary Disease (COPD) are locked in a vicious circle of inactivity and social isolation which profoundly affects their quality of life and prognosis. A new wearable non invasive positive pressure ventilation device has been recently proposed; it can be used by intermittence during or after physical activities for reducing dyspnea or for shortening dyspnea- recovery time. The investigators hypothesize that this system, in reducing the inconvenience caused by dyspnea, would stimulate a more active lifestyle and improve quality of life. Their objective is to assess the impact of this device on physical activity and quality of life in patients with severe COPD, complaining of dyspnea.

In this open study with no control group, participants will use the device at their convenience, according to their needs in daily life and for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable severe COPD (with FEV1 ≤50% predicted)
* Patients with mMRC score > ou = 2.

Exclusion Criteria:

* Exacerbate within a month prior.
* Using other non invasive ventilation device > 15h per day.
* Have musculoskeletal or neuromuscular problem affecting balance and walking.
* Have cognitive problem affecting comprehension of the different évaluations or questionnaires.
* Have recently participated in physical training or rehabilitation program (≤ 3 months).
* Medical contra-indication to NIV.
* Evolutionary pathologies (excluding COPD) may be life-threatening in the short term (1 year) (cancer, neuromuscular disease rapidly changing).
* Simultaneously enrolled in an other clinical trial.
* Not affiliated to social security.
* Person deprived of liberty, major protected by law.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Change of daily physical activity measured by actimetry | Continuously over a 8-week period (2 weeks before the use of the device, over the 4-week period usinf the device and 2 weeks after the use of the device
  Change of number of steps by day and daily energy expenditure over the 8 week period

SECONDARY OUTCOMES:
Change of Baseline Dyspnea Index (BDI) score | baseline and post use of the Vitabreath device at 4th weeks
  The BDI represents importance and impact of dyspnea in daily life of COPD patients. The BDI is one of dyspnea parameters (questionnaire). Three dimension questions include; 1.effect of daily function on dyspnea, 2. effect of magnitude of task on dyspnea and 3. effect of magnitude off effort on dyspnea.
Change of Modified Medical Research Council Questionnaire (mMRC) score | baseline and post use of the Vitabreath device at 4th weeks
  The mMRC is one of dyspnea parameters
Change of Transition Dyspnea Index (TDI) | baseline and post use of the Vitabreath device at 4th weeks
  The TDI assesses change of dyspnea perception from the BDI in each dimensions. Patient will rate score from -6 to +6 (positive score reflect improve of dyspnea and negative score reflect worse dyspnea).
Subjective appréciation of the device | post use of the Vitabreath device at 4th weeks
  Patients will rate their appreciation of the device using 3 scale relatives to ease of use, helps recovery shortness of breath, helps to be more active in daily life
Change of Visual Simplified Respiratory Questionnaire (VSRQ) score | baseline and post use of the Vitabreath device at 4th weeks
  The VRSQ represents health related quality of life of COPD patients
Change of Chronic Obstructive Pulmonary Disease Assessment Test (CAT)score | Continuously over a 8-week period (2 weeks before the use of the device, over the 4-week period usinf the device and 2 weeks after the use of the device
  The CAT represents health related quality of life of COPD patients

OTHER OUTCOMES:
Compliance to the device | Every week over the 4-week period
  During a weekly phone call, patients will indicate the daily duration and conditions of use of the device
Number of acute exacerbation | Up to 12 months before the date of inclusion
  Exacerbation is defined as changing the respiratory status of the patient relative to the patient's usual state, which requires acute hospitalisation.
Weight | baseline and post use of the Vitabreath device at 4th weeks
  Patient will indicate their weight

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, Pr, Principal Investigator — Laboratoire du sommeil - Centre hospitalier Universitaire Michallon - 38043 GRENOBLE
Locations (7):
- France (7):
  - Dr Michèle Bognie Pneumology Office, Alès
  - Clinique du Parc, Castelnau-le-Lez
  - CHU Grenoble-Alpes, Grenoble
  - Hôpital Privé La Louvière, Lille
  - Dr Christian PAILLARGUELO Pneumology Office, Lunel
  - CHU Caremeau, Nîmes
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided